CLINICAL TRIAL: NCT01586442
Title: A Comparison of the Effects of Selective and Non Selective Mineralocorticoid Antagonism on Glucose Homeostasis and Lipid Profile of Heart Failure Patients With Glucose Intolerance or Type 2 Diabetes.
Brief Title: Comparison of Eplerenone Versus Spironolactone in Heart Failure Patients With Glucose Intolerance or Type 2 Diabetes
Acronym: SNOW
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Michel White, Michel White, MD, FRCP(C), FACC, FESC, Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WS1911307
Record Dates: First submitted 2012-04-24; First posted 2012-04-26 (Estimated); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure; Type 2 Diabetes; Glucose Intolerance
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus, Type 2; Glucose Intolerance | interventions — Eplerenone; Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spironolactone (Active Comparator): spironolactone 12.5mg once daily titrated to 25mg once daily
  Interventions: Drug: Spironolactone
- Eplerenone (Experimental): Eplerenone 25mg once daily titrated to 50mg once daily
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone — Eplerenone 25mg once daily titrated to 50 mg once daily for 4 months
  Other Names: Inspra
  Arms: Eplerenone
Drug: Spironolactone — Spironolactone 12,5mg daily titrated to 25mg once daily for 16 weeks
  Other Names: Aldactone
  Arms: Spironolactone

SUMMARY:
In this proposal,the investigators will examine whether the selectivity of eplerenone for the MR will translate into a better glucose and metabolic profile compare to spironolactone in patients with HF with glucose intolerance or type 2 diabetes. In addition, the investigators will also compare the impact of these two agents on changes of concentrations of established prognostic biomarkers of neurohormonal activation and extracellular matrix turnover.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 18 years old.
2. Symptomatic HF corresponding to NYHA class II-IV symptoms for at least 4 weeks prior randomization.
3. A diagnosis of 1) impaired glucose tolerance described as overnight fasting between blood glucose 5.6 and 6.9 mmol/L on two occasions; or 2) type 2 diabetes defined as overnight fasting between blood glucose of 7.0 mmol/L or more on two occasions; a HbA1c equal to or higher than 6.5% or more on two occasions; or as a history of type II diabetes treated with hypoglycemic agents.
4. LVEF equal to or lower than 40% documented by, contrast ventriculography, magnetic resonance imaging, radionuclide ventriculography or quantitative echocardiography within the previous 12 months if no cardiac event occurred since the measurement of the LVEF. The most recent measurements should be used.
5. Treatment with an optimal and stable dose of ACE inhibitor (or ARB) for at least 4 weeks prior to enrolment in the study. In addition, patients should be treated with a stable dose of beta-blockers for at least 4 weeks prior enrolment in the study. Patients incapable to tolerate bisoprolol, carvedilol or metoprolol will be allowed within the trial.
6. Informed consent must be obtained before any study specific procedures are performed

Exclusion Criteria:

1. Current treatment with a combination of an ARB, an ACE or a renin inhibitor.
2. Type 1 diabetes
3. Known intolerance or allergy to eplerenone or spironolactone, including gynecomastia with spironolactone.
4. Estimated GFR < 30 mL/min/1.73 m2 as calculated using the MDRD equation (Appendix 1).
5. Current serum potassium higher than 5.0 mmol/L (higher than 5.0 mEq/L).
6. Current symptomatic hypotension and/or systolic B.P. < 90 mmHg.
7. Persistent systolic or diastolic hypertension (systolic > 170 mmHg or diastolic > 100 mmHg despite use of antihypertensive therapy).
8. HF secondary to any of the following conditions: hemodynamically significant primary stenotic valvular cardiomyopathy, isolated right sided CHF, non cardiac disease (e.g. uncorrected thyroid disease), pericardial disease, complex congenital heart disease, myocarditis.
9. Decompensated heart failure described as hospitalization or I.V. administration of medication in emergency room or heart failure clinic within 4 weeks (ex.: diuretics, inotropes, vasodilatators)
10. Current treatment with insulin
11. Stroke, acute coronary syndrome, PCI within the last 4 weeks before randomization.
12. Cardiac surgery within 3 months.
13. Significant liver disease (ALT x 3 times limit of normal).
14. Planned cardiac surgery expected to be performed within the next 6 months.
15. Previous heart transplant or heart transplant expected to be performed within the next 6 months.
16. Presence of any non-cardiac diseases likely to significantly shorten life expectancy to < 1 year.
17. Pregnant or lactating women or women of childbearing potential who are not protected from pregnancy by an accepted method of contraception, such as the oral contraceptive pill, an intrauterine device or surgical sterilization (all women of childbearing potential must have a negative pregnancy test before randomization).
18. Any condition that in the opinion of the investigator would jeopardize the evaluation on efficacy or safety or be associated with poor adherence to the protocol.
19. Treatment with any investigational agent or device within 4 weeks of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-03; Primary Completion 2015-03 (Actual); Study Completion 2018-07-29 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin | 4 months
  Change in glycated hemoglobin
Fasting glucose and lipid profile | 4 months
Plasma insulin | 4 months
Cortisol | 4 months
Adiponectin | 4 months
NT-proBNP | 4 months
PIIINP | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Michel White, MD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Korol S, White M, O'Meara E, Tournoux F, Racine N, Ducharme A, Rouleau JL, Liszkowski M, Mansour A, Jutras M, Guertin MC, Bernier M, Lavoie J, Leclair G, Neagoe PE, Chaar D, Sirois MG, de Denus S. A comparison of the effects of selective and non-selective mineralocorticoid antagonism on glucose homeostasis of heart failure patients with glucose intolerance or type II diabetes: A randomized controlled double-blind trial. Am Heart J. 2018 Oct;204:190-195. doi: 10.1016/j.ahj.2018.07.002. Epub 2018 Jul 10. PMID 30097164